CLINICAL TRIAL: NCT01241890
Title: Prevention of CF Exacerbation in Childhood (PREVEC): Early Recognition of Inflammation by Non-invasive Biomarkers in Exhaled Breath (Condensate)
Brief Title: Prevention of CF Exacerbation in Childhood: PREVEC Study
Acronym: PREVEC
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: NCFS (Unknown); Chiesie Pharmaceuticals B.V. (Unknown)
Responsible Party: Sponsor
Other Study IDs: MEC 11-3-111
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Cystic Fibrosis; Children; Exhaled Breath Condensate; Non-invasive Inflammatory Markers; Volatile Organic Compounds; Home Monitoring; Quality of Life
Keywords: Cystic Fibrosis; Children; Exhaled Breath Condensate; Non-invasive Inflammatory Markers; Volatile Organic Compounds; Home monitoring; Quality of life
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children with Cystic Fibrosis, care as usual: Treatment according to the Dutch Central Guidance Committee (CBO) guidelines for CF. Assessments: home monitoring, symptoms, lung function, quality of life and diagnostic assessments of non-invasive inflammatory markers in exhaled air and exhaled breath condensate.

SUMMARY:
Pulmonary exacerbations of CF are an important cause for the experienced disability of patients, respiratory symptoms, and decreases in lungfunction, which require antibiotic therapy at home or in the hospital. Therefore, prevention of exacerbations in CF is important. The aim of this study was to assess the predictive properties of inflammatory markers in exhaled breath for pulmonary exacerbations in children with CF. In addition the reliability of home monitor assessments of symptoms and lungfunction was investigated.

ELIGIBILITY:
Inclusion Criteria:

* CF disease is defined as the combination of:

  1. characteristic clinical features (persistent pulmonary symptoms, meconium ileus, failure to thrive, steatorrhoea);
  2. and/or abnormal sweat test (Chloride > 60mM);
  3. and/or two CF mutations.

Exclusion Criteria:

1. cardiac abnormalities;
2. mental retardation;
3. no technical satisfactory performance of measurements;
4. on the waiting list for lung transplantation;
5. non-compliance with the home-assessments;
6. patients with Burkholderia Cepacia;
7. participation in another intervention trial.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with Cystic Fibrosis
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2011-10; Primary Completion 2013-08 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Number of exacerbations | 1 year
  Definition of an exacerbation according to Treggiari MM et al.

SECONDARY OUTCOMES:
Quality of life | 1 year
  Quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: E Dompeling, PhD MD, Principal Investigator — Maastricht University Medical Centre
Locations (3):
- Netherlands (3):
  - Academic Medical Centre, Amsterdam
  - Maastricht University Medical Centre, Maastricht
  - University Medical Centre, Utrecht